CLINICAL TRIAL: NCT03008486
Title: Long Term Effects of Soft Splints on Stroke Patients and Patients With Disorders of Consciousness
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Géraldine Martens (Other)
Collaborators: Centre Hospitalier Universitaire UCLouvain Namur (Other)
Responsible Party: Sponsor-Investigator, Géraldine Martens, PhD student, University of Liege
Organization: University of Liege (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2016/292
Record Dates: First submitted 2016-12-26; First posted 2017-01-02 (Estimated); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Brain Injuries; Disorder of Consciousness; Stroke; Spasticity as Sequela of Stroke; Contracture; Hypertonic Disorder; Central Nervous System Diseases; Pathologic Processes; Craniocerebral Trauma; Trauma, Nervous System; Neurocognitive Disorders
MeSH Terms: conditions — Brain Injuries; Consciousness Disorders; Stroke; Contracture; Central Nervous System Diseases; Pathologic Processes; Craniocerebral Trauma; Trauma, Nervous System; Neurocognitive Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- DOC - real (Active Comparator): Spastic patients with disorders of consciousness receiving the real soft splint
  Interventions: Device: Real soft splint (6 cm)
- DOC - placebo (Placebo Comparator): Spastic patients with disorders of consciousness receiving the placebo soft splint
  Interventions: Device: Placebo soft splint (1 cm)
- Stroke - real (Active Comparator): Spastic patients stroke receiving the real soft splint
  Interventions: Device: Real soft splint (6 cm)
- Stroke - placebo (Placebo Comparator): Spastic patients stroke receiving the placebo soft splint
  Interventions: Device: Placebo soft splint (1 cm)

INTERVENTIONS:
Device: Real soft splint (6 cm)
  Arms: DOC - real; Stroke - real
Device: Placebo soft splint (1 cm)
  Arms: DOC - placebo; Stroke - placebo

SUMMARY:
The purpose of this study is to assess the effects on upper limb spasticity of soft splints worn during three weeks three hours a day by patients with stroke or disorders of consciousness.

DETAILED DESCRIPTION:
Patients with stroke or disorders of consciousness (DOC) are likely to suffer from major muscular troubles such as spasticity. This spasticity may induce pain, loss in range of motion and permanent joint deformities. The aim of this study is to investigate the effects of soft splinting on the hand spasticity in both patients with stroke and patients with disorders of consciousness. The investigators plan to include 100 patients (50 stroke - 50 with DOC) and each subgroup will be divided in two arms: one wearing real soft splints (6 cm diameter) three hours a day for 3 three weeks and the other one wearing 'placebo' splints (1 cm diameter).

Skin condition will be followed by the nursing team during the three weeks. Spasticity, pain and consciousness assessments will be performed at baseline (week 0), after 1 week of treatment (week 1) at the end of the treatment (week 3), 1 week later (week 4), 3 weeks later (week 6) and three months later (week 12).

ELIGIBILITY:
Inclusion Criteria (DOC):

* Altered state of consciousness according to international criteria since more than three months
* Stable condition
* Ashworth score > 1 for at least one upper limb joint

Exclusion Criteria:

* Bone fracture/lesion at the upper limbs
* Serious neurological disorder (MMSE > 24) prior to the accident
* Botox injection on the upper limbs in the 6 months preceding the inclusion

Inclusion Criteria (stroke):

* Central nervous system injury responsible for the spasticity
* Ashworth score > 1 for at least one upper limb joint

Exclusion Criteria:

* Bone fracture/lesion at the upper limbs
* Serious neurological disorder (MMSE > 24)
* Botox injection on the upper limbs in the 6 months preceding the inclusion

Ages: 14 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2017-01; Primary Completion 2019-01 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
Change in the Modified Ashworth Scale | Week 0, 1, 3, 4, 6, 12
  Spasticity assessment
Change in the Modified Tardieu Scale | Week 0, 1, 3, 4, 6, 12
  Spasticity assessment
Change in the Nociception Coma Scale-Revised | Week 0, 1, 3, 4, 6, 12
  Pain assessment
Change in the Visual Analogue Scale | Week 0, 1, 3, 4, 6, 12
  Pain assessment
Change in the Palm-finger distance | Week 0, 1, 3, 4, 6, 12
  Range of motion assessment

SECONDARY OUTCOMES:
Change in the Coma Recovery Scale-Revised | Week 0, 1, 3, 4, 6, 12
  Consciousness assessment

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Lejeune, Principal Investigator — Centre Hospitalier Neurologique William Lennox
Locations (1):
- Centre Hospitalier Neurologique William Lennox, Ottignies, Brabant Wallon, Belgium

IPD SHARING:
Plan to Share IPD: No